CLINICAL TRIAL: NCT03667040
Title: A Randomized Controlled Trial of an E-health Resilience Program For Chronic Spine Pain
Brief Title: E-health Resilience Program For Chronic Spine Pain
Acronym: JOOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Afton Hassett, Psy.D., Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00146178
Record Dates: First submitted 2018-09-07; First posted 2018-09-12 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Back Pain; Neck Pain
MeSH Terms: conditions — Back Pain; Neck Pain

STUDY DESIGN:
Intervention Model Description: 150 participants will be recruited; 75 participants into the intervention group and 75 into the control group. There will three visits, baseline and follow-up at 30 days and 60 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): 75 participants will take part in three visits (baseline, 30days and 60days)
- Intervention (Active Comparator): 75 participants will take complete a baseline visit and then participate in the intervention. They will use the application, the JOOL app for 30 days. Then complete surveys at 30days and 60days after the interventions
  Interventions: Behavioral: JOOL app

INTERVENTIONS:
Behavioral: JOOL app — Participants will use the JOOL app for 30 days
  Arms: Intervention

SUMMARY:
This study will examine a e-health resilience based program, JOOL, for chronic spine pain patients through the following aims:

Aim 1: To test the effectiveness of a resilience based program known as JOOL Aim 2: To evaluate the characteristics of the participants most likely to benefit from this treatment

DETAILED DESCRIPTION:
This is a pilot RCT in which 150 patients with chronic spine pain will be randomized to one of two arms: (1) a group that downloads the JOOL mobile application resilience program; and (2) a control group.The primary outcome will be a change in physical function.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the UM Back & Pain Center
* Primary diagnosis of neck or back pain (spine pain)
* Age 18-70
* English speaking
* Able to provide consent
* Willing to download the mobile application and comply with study procedures
* Antidepressant medications stable for ≥ 4 weeks
* No plan to initiate a new non-pharmacological pain intervention during the 30-day study period (e.g. back surgery, physical therapy, behavioral therapy

Exclusion Criteria

* Having known psychotic disorder or the presence of another psychiatric condition (e.g. severe depression [HADS scores ≥ 15], suicidal ideation) or cognitive impairment (e.g. severe dyslexia, TBI) limiting ability to give consent and/or participate fully in the study
* Currently undergoing psychotherapeutic care at the Back & Pain Center because many of the concepts that are the focus of this study are already employed in that treatment
* Other factors that at the discretion of the investigators would adversely affect study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
PROMIS (Patient Reported Outcomes Measurement Information System) Physical Function Scale- Short form 10 | 2 month
  10 item survey measuring physical function. Each question is measured on a scale of 1-5. The lowest score being 10 and highest score is 50. A higher score correlates with poor physical functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Afton Hassett, PsyD, Principal Investigator — University of Michigan
Locations (1):
- Back & Pain Center, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided